CLINICAL TRIAL: NCT00005763
Title: INTERSALT: International Study of Sodium, Potassium, and Blood Pressure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Wellcome Trust (Other)
Other Study IDs: 1045; R01HL033387 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To coordinate an international study on the relationships between population mean sodium and potassium intake and blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

For decades diet, particularly high habitual sodium intake, has been implicated in the etiopathogenesis of high blood pressure. This concept has been based on clinical observations, including therapeutics and results of dietary trials; on animal experimentation, particularly induction of hypertension by salt feeding; and on epidemiologic findings. While considerable knowledge has been amassed in support of this concept, limitations and inconsistencies exist in the data base. This is especially true in regard to the findings from population studies. Thus, negative or inconsistent results have been reported from several cross-sectional studies of dietary sodium and blood pressure in which the unit of measurement has been the individual within a population. When INTERSALT began in 1984, no prospective data were available from population-based longitudinal investigations. A major problem in such studies, one possibly accounting for the negative and inconsistent findings, was the difficulty of validly measuring the habitual sodium intake of individuals within a population in which there was relative homogeneity in regard to this trait. This difficulty was due to large individual variation day-to-day in the sodium intake and output in most populations, so that the ratio of intra- to inter-individual variances was large. This led to high probability of misclassification and obscuring or weakening of true associations in any single population sample, unless multiple measurements were made for each person. Since dietary history methods such as 7-day food records, multiple 24-hour recalls, and dietary interviews were of limited validity for assessment of sodium intake, investigators had to rely on timed urine collections, especially 24-hour samples. But accurate collection of several such specimens per person by many individuals for population studies was a difficult undertaking. This was an important reason for the paucity of valid data on sodium and blood pressure from within-population studies.

INTERSALT was based on a common protocol and had a staff trained in standardized procedures in each center, thus permitting estimation of the sodium-blood pressure relationship within as well as across centers. INTERSALT originated as a Project of the Council on Epidemiology and Prevention of the International Society and Federation of Cardiology and has since its inception been jointly coordinated by the London School of Hygiene and Tropical Medicine and the Northwestern University Medical School. The main data analyses were performed in London. Overwhelmingly, funding for the work of the London Coordinating Center, the Central Laboratory, as well as for the 52 centers, had been organized independently. For example, support came from the Wellcome Trust, the World Health Organization, the International Society of Hypertension, the Council on Epidemiology and Prevention of the International Society and Federation of Cardiology, the Dutch Heart Foundation, the British Heart Foundation, the Canadian Heart Foundation, the Japanese Heart Foundation, as well as the private sector.

The grant to Northwestern University supported the Chicago share of training and coordination of the Chicago population sample of the Peoples Gas Company, assistance to six centers in developing countries, part of the Coordinating Center and the Central Laboratory, and some of the data analysis. The grant to the University of Mississippi supported the four population samples in Mississippi.

DESIGN NARRATIVE:

A common protocol was followed in this cross-sectional study. Data were collected on blood pressure and on electrolyte and creatinine excretion in timed 24-hour urine and casual urine samples. Data were also collected on age, sex, height, weight, alcohol intake, diet, drug treatment for hypertension, family history of cardiovascular disease, contraceptive pill use, smoking, physical activity, and social and educational status. Urine specimens were analyzed for sodium, potassium, chloride, calcium, magnesium, and creatinine in the central laboratory at St. Raphael University in Leuven, Belgium. The data were coordinated at the London School of Hygiene and Tropical Medicine, London, England. The data from the University of Mississippi were analyzed separately using uric acid as a covariate.

The study was renewed in 1992 to conduct further analysis. Based on the important findings of an inverse association between urinary markers of protein intake and blood pressure in analyses conducted on 12 of the 52 INTERSALT centers, the first component of the renewal study was to complete the biochemical and statistical analyses for the 52 centers and provide the first large population-based assessment to test the hypothesis of an inverse relationship of dietary protein to BP of individuals (with N=10,079). This relationship was also examined across populations having a wide variety of nutritional patterns (N = 52). The second major component of the study renewal was to assess the impact protein intake had on the original INTERSALT findings of a significant relation of Na, K, and Na/K with blood pressure. This component included investigation of possible interactions of Na, K, and Na/K with protein as well as with other factors shown in INTERSALT to relate to blood pressure. In addition to these main substantive questions, methodologic issues related to assessment of nutritional factors and blood pressure were further investigated.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1984-12; Study Completion 1997-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Stamler

REFERENCES:
- [Background] Elliott P, Stamler J, Nichols R, Dyer AR, Stamler R, Kesteloot H, Marmot M. Intersalt revisited: further analyses of 24 hour sodium excretion and blood pressure within and across populations. Intersalt Cooperative Research Group. BMJ. 1996 May 18;312(7041):1249-53. doi: 10.1136/bmj.312.7041.1249. PMID 8634612
- [Background] Hanneman RL. Intersalt: hypertension rise with age revisited. BMJ. 1996 May 18;312(7041):1283-4; discussion 1284-7. doi: 10.1136/bmj.312.7041.1283. No abstract available. PMID 8634620
- [Background] Law M: Commentary: Evidence on Salt is Consistent. (Not supported by the grant. This is another commentary.) BMJ, 312:1284-1285, 1996
- [Background] Dyer AR, Elliott P, Marmot M, Kesteloot H, Stamler R, Stamler J. Commentary: strength and importance of the relation of dietary salt to blood pressure. Intersalt Steering and Editorial Committee. BMJ. 1996 Jun 29;312(7047):1661-4. doi: 10.1136/bmj.312.7047.1661. No abstract available. PMID 8664726
- [Background] Naruse Y, Nakagawa H, Kagamimori S, Fujita Y, Hashimoto T, Kasamatsu T, Mikawa K, Ueshima H. Relationship of parental history of high blood pressure to blood pressure: combined findings of three Japanese population samples, the INTERSALT study. J Hum Hypertens. 1998 Apr;12(4):215-20. doi: 10.1038/sj.jhh.1000469. PMID 9607688
- [Background] Rennolls K. Intersalt data. Science demands data sharing. BMJ. 1997 Aug 23;315(7106):486-7. No abstract available. PMID 9284679
- [Background] Liebman BF, Jacobson MF. Intersalt data. Sodium contents of restaurant foods in United States are high. BMJ. 1997 Aug 23;315(7106):488. No abstract available. PMID 9284681
- [Background] Grimm RH. Intersalt data. Collaborative efforts must be made to reduce sodium in diet. BMJ. 1997 Aug 23;315(7106):487. No abstract available. PMID 9284680
- [Background] Davey Smith G, Phillips AN. Intersalt data. Correction for regression dilution bias in Intersalt study was misleading. BMJ. 1997 Aug 23;315(7106):485-6; author reply 487. No abstract available. PMID 9284677
- [Background] Day NE. Intersalt data. Epidemiological studies should be designed to reduce correction needed for measurement error to a minimum. BMJ. 1997 Aug 23;315(7106):485; author reply 487. No abstract available. PMID 9284676
- [Background] Macnair A. Intersalt data. Conclusions drawn in paper "revisiting" Intersalt data are of questionable validity. BMJ. 1997 Aug 23;315(7106):485; author reply 487. No abstract available. PMID 9284675
- [Background] Alderman M. Intersalt data. Data linking sodium intake to subsequent morbid and fatal outcomes must be studied. BMJ. 1997 Aug 23;315(7106):484-5; author reply 487. No abstract available. PMID 9284674
- [Background] Dyer A, Elliott P, Chee D, Stamler J. Urinary biochemical markers of dietary intake in the INTERSALT study. Am J Clin Nutr. 1997 Apr;65(4 Suppl):1246S-1253S. doi: 10.1093/ajcn/65.4.1246S. PMID 9094929
- [Background] Stamler J, Elliott P, Kesteloot H, Nichols R, Claeys G, Dyer AR, Stamler R. Inverse relation of dietary protein markers with blood pressure. Findings for 10,020 men and women in the INTERSALT Study. INTERSALT Cooperative Research Group. INTERnational study of SALT and blood pressure. Circulation. 1996 Oct 1;94(7):1629-34. doi: 10.1161/01.cir.94.7.1629. PMID 8840854
- [Background] Joossens JV, Hill MJ, Elliott P, Stamler R, Lesaffre E, Dyer A, Nichols R, Kesteloot H. Dietary salt, nitrate and stomach cancer mortality in 24 countries. European Cancer Prevention (ECP) and the INTERSALT Cooperative Research Group. Int J Epidemiol. 1996 Jun;25(3):494-504. doi: 10.1093/ije/25.3.494. PMID 8671549
- [Background] INTERSALT Study an international co-operative study on the relation of blood pressure to electrolyte excretion in populations. I. Design and methods. The INTERSALT Co-operative Research Group. J Hypertens. 1986 Dec;4(6):781-7. doi: 10.1097/00004872-198612000-00014. PMID 3819392
- [Background] Elliott P, Stamler R. Manual of operations for "INTERSALT", an international cooperative study on the relation of sodium and potassium to blood pressure. Control Clin Trials. 1988 Jun;9(2 Suppl):1S-117S. No abstract available. PMID 3396367
- [Background] Intersalt: an international study of electrolyte excretion and blood pressure. Results for 24 hour urinary sodium and potassium excretion. Intersalt Cooperative Research Group. BMJ. 1988 Jul 30;297(6644):319-28. doi: 10.1136/bmj.297.6644.319. PMID 3416162
- [Background] Stamler J, Rose G, Stamler R, Elliott P, Dyer A, Marmot M. INTERSALT study findings. Public health and medical care implications. Hypertension. 1989 Nov;14(5):570-7. doi: 10.1161/01.hyp.14.5.570. PMID 2807518
- [Background] Rose G, Stamler J. The INTERSALT study: background, methods and main results. INTERSALT Co-operative Research Group. J Hum Hypertens. 1989 Oct;3(5):283-8. PMID 2810325
- [Background] Elliott P, Marmot M, Dyer A, Joossens J, Kesteloot H, Stamler R, Stamler J, Rose G. The INTERSALT study: main results, conclusions and some implications. Clin Exp Hypertens A. 1989;11(5-6):1025-34. doi: 10.3109/10641968909035389. PMID 2791323
- [Background] Elliott P, Dyer A, Stamler R. The INTERSALT study: results for 24 hour sodium and potassium, by age and sex. INTERSALT Co-operative Research Group. J Hum Hypertens. 1989 Oct;3(5):323-30. PMID 2810328
- [Background] Dyer AR, Elliott P. The INTERSALT study: relations of body mass index to blood pressure. INTERSALT Co-operative Research Group. J Hum Hypertens. 1989 Oct;3(5):299-308. PMID 2810326
- [Background] Elliott P. The INTERSALT study: an addition to the evidence on salt and blood pressure, and some implications. J Hum Hypertens. 1989 Oct;3(5):289-98. PMID 2681780
- [Background] Carvalho JJ, Baruzzi RG, Howard PF, Poulter N, Alpers MP, Franco LJ, Marcopito LF, Spooner VJ, Dyer AR, Elliott P, et al. Blood pressure in four remote populations in the INTERSALT Study. Hypertension. 1989 Sep;14(3):238-46. doi: 10.1161/01.hyp.14.3.238. PMID 2767757
- [Background] Dyer AR, Elliott P, Shipley M. Body mass index versus height and weight in relation to blood pressure. Findings for the 10,079 persons in the INTERSALT Study. Am J Epidemiol. 1990 Apr;131(4):589-96. doi: 10.1093/oxfordjournals.aje.a115543. PMID 2180281
- [Background] Elliott P, Rogers S, Scally G, Beevers DG, Lichtenstein MJ, Keenan G, Hornby R, Evans A, Shipley MJ, Elwood PC. Sodium, potassium, body mass, alcohol and blood pressure in three United Kingdom centres (the INTERSALT study). Eur J Clin Nutr. 1990 Sep;44(9):637-45. PMID 2261896
- [Background] Stamler J, Rose G, Elliott P, Dyer A, Marmot M, Kesteloot H, Stamler R. Findings of the International Cooperative INTERSALT Study. Hypertension. 1991 Jan;17(1 Suppl):I9-15. doi: 10.1161/01.hyp.17.1_suppl.i9. PMID 1987018
- [Background] Stamler R. Implications of the INTERSALT study. Hypertension. 1991 Jan;17(1 Suppl):I16-20. doi: 10.1161/01.hyp.17.1_suppl.i16. No abstract available. PMID 1986996
- [Background] Stamler R, Shipley M, Elliott P, Dyer A, Sans S, Stamler J. Higher blood pressure in adults with less education. Some explanations from INTERSALT. Hypertension. 1992 Mar;19(3):237-41. doi: 10.1161/01.hyp.19.3.237. PMID 1548050
- [Background] Marmot MG, Elliott P, Shipley MJ, Dyer AR, Ueshima H, Beevers DG, Stamler R, Kesteloot H, Rose G, Stamler J. Alcohol and blood pressure: the INTERSALT study. BMJ. 1994 May 14;308(6939):1263-7. doi: 10.1136/bmj.308.6939.1263. PMID 7802765
- [Background] Dyer AR, Elliott P, Shipley M, Stamler R, Stamler J. Body mass index and associations of sodium and potassium with blood pressure in INTERSALT. Hypertension. 1994 Jun;23(6 Pt 1):729-36. doi: 10.1161/01.hyp.23.6.729. PMID 8206570
- [Background] Le Fanu J. Intersalt data. Cross cultural studies such as Intersalt study cannot be used to infer causality. BMJ. 1997 Aug 23;315(7106):484; author reply 487. No abstract available. PMID 9284673
- [Background] Watt G, Hart JT. Intersalt data. Slow decremental change in dietary sodium load in whole populations is needed. BMJ. 1997 Aug 23;315(7106):486; author reply 487. No abstract available. PMID 9284678
- [Background] Stamler J. The INTERSALT Study: background, methods, findings, and implications. Am J Clin Nutr. 1997 Feb;65(2 Suppl):626S-642S. doi: 10.1093/ajcn/65.2.626S. PMID 9022559
- [Background] Elliott P, Dyer A, Stamler R, Stamler J. Correcting for regression dilution in INTERSALT. Lancet. 1993 Oct 30;342(8879):1123. doi: 10.1016/0140-6736(93)92112-7. No abstract available. PMID 8105352